CLINICAL TRIAL: NCT04713930
Title: A Randomized, Placebo-controlled, Double-blind, Single Ascending Dose Study to Investigate Safety, Tolerability, and Pharmacokinetics of JNJ-61393215 in Healthy Japanese Adult Male Subjects
Brief Title: A Study of JNJ-61393215 in Healthy Japanese Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: CR108937; 61393215EDI1005 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2021-01-15; First posted 2021-01-19 (Actual); Last update posted 2025-04-28 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — Hcrtr1 protein, mouse

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JNJ-61393215 (Experimental): Participants will receive one of 3 single oral doses of JNJ-61393215 on Day 1, escalated sequentially based on the safety review in Cohorts 1, 2, and 3 up to Day 5.
  Interventions: Drug: JNJ-61393215
- Placebo (Active Comparator): Participants will receive a single oral dose of placebo on Day 1 in Cohorts 1, 2, and 3 up to Day 5.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-61393215 — JNJ-61393215 will be administered orally.
  Other Names: Orexin-1
  Arms: JNJ-61393215
Drug: Placebo — Placebo will be administered orally.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (PK) after single dose administrations of JNJ-61393215 in Japanese healthy adult male participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI = weight/height^2) between 18 and 30 kilogram per meter square (kg/m^2) (inclusive), and body weight not less than 50 kilogram (kg)
* Be healthy on the basis of physical examination, medical history, vital signs, and 12 lead electrocardiogram (ECG) (including QT interval corrected according to Fridericia's formula [QTcF] less than or equal to [<=] 450 millisecond [msec]) performed at screening. Minor abnormalities in ECG, which are not considered to be of clinical significance by the investigator, are acceptable
* Healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Blood pressure (after the participant supine for at least 5 minutes) 90 millimeter of Mercury (mmHg) or more and less than 140 mmHg systolic, and less than 90 mmHg diastolic. If blood pressure is out of range, up to 2 repeated assessments are permitted
* During the study and for a minimum of one spermatogenesis cycle (defined as approximately 90 days) after receiving (the last dose of) study intervention, in addition to the highly effective method of contraception, a man a) who is sexually active with a woman of childbearing potential must agree to use a barrier method of contraception (example, condom with spermicidal foam/gel/film/cream/suppository), b) who is sexually active with a woman who is pregnant must use a condom, c) must agree not to donate sperm. In addition, recommended highly effective methods of contraception in this study for female partners of male participants to use in addition to the male participant wearing a condom include: a) oral hormonal contraception, b) intrauterine device, c) intrauterine hormone-releasing system, and d) bilateral tubal occlusion

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening as deemed appropriate by the investigator
* Clinically significant abnormal physical examination, vital signs, or 12 lead ECG at screening as deemed appropriate by the investigator
* Known allergies, hypersensitivity, or intolerance to JNJ-61393215 or its excipients
* Test positive for human immunodeficiency virus (HIV) antigen/antibodies, hepatitis A antibody immunoglobulin M (IgM), syphilis, hepatitis B surface antigen (HbsAg) or hepatitis C virus (HCV) antibodies at screening

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 42 days
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Plasma Concentration of JNJ-61393215 | Predose, up to 96 hours postdose (up to Day 5)
  Plasma samples will be analyzed to determine concentrations of JNJ-61393215 using a validated, specific, and sensitive liquid chromatography mass spectrometry/mass spectrometry (LC-MS/MS).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Souseikai Hakata Clinic, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinicaltrials/ transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency